CLINICAL TRIAL: NCT03347123
Title: A Phase 1/2, Open-Label, Dose-Escalation, Safety, Tolerability, and Efficacy Study of Epacadostat and Nivolumab in Combination With Immune Therapies in Subjects With Advanced or Metastatic Malignancies (ECHO-208)
Brief Title: A Study of Epacadostat and Nivolumab in Combination With Immune Therapies in Participants With Advanced or Metastatic Malignancies (ECHO-208)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A business decision made by Incyte after analysis of data from a sister study.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 24360-208 (ECHO-208); 2017-001743-12 (EudraCT Number)
Record Dates: First submitted 2017-11-14; First posted 2017-11-20 (Actual); Results first posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Solid Tumors
Keywords: Epacadostat; nivolumab; ipilimumab; lirilumab; solid tumor; melanoma; non-small cell lung cancer (NSCLC); squamous cell carcinoma of the head and neck (SCCHN); IDO inhibitor
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — epacadostat; Nivolumab; Ipilimumab; lirilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1: Dose Escalation: Treatment Group A: Cohort 1 Epacadostat 50 mg BID (Experimental): Participants with advanced or metastatic solid tumor who have received no more than 2 prior treatment regimens received epacadostat 50 mg BID orally in combination with nivolumab 240 mg on day 1 of each 14 day cycle and ipilimumab 1 mg/kg intravenous (IV) every 6 weeks thereafter on Day 1 of every third treatment cycle until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 24 months.
  Interventions: Drug: Epacadostat; Drug: Nivolumab; Drug: Ipilimumab
- Phase 1: Dose Escalation: Treatment Group A: Cohort 2 Epacadostat 100 mg BID (Experimental): Participants with advanced or metastatic solid tumor who have received no more than 2 prior treatment regimens received epacadostat 100 mg BID orally in combination with nivolumab 240 mg on day 1 of each 14 day cycle and ipilimumab 1 mg/kg intravenous (IV) every 6 weeks thereafter on Day 1 of every third treatment cycle until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 24 months.
  Interventions: Drug: Epacadostat; Drug: Nivolumab; Drug: Ipilimumab
- Phase 1: Dose Escalation: Treatment Group B: Cohort 1 Epacadostat 50 mg BID (Experimental): Participants with advanced or metastatic solid tumor who have received no more than 2 prior treatment regimens received epacadostat 50 mg BID orally in combination with nivolumab 240 mg on day 1 of every 14 day cycle and lirilumab 240 mg IV every 4 weeks until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 24 months.
  Interventions: Drug: Epacadostat; Drug: Nivolumab; Drug: Lirilumab
- Phase 1: Dose Escalation: Treatment Group B: Cohort 2 Epacadostat 100 mg BID (Experimental): Participants with advanced or metastatic solid tumor who have received no more than 2 prior treatment regimens received epacadostat 100 mg BID orally in combination with nivolumab 240 mg on day 1 of every 14 day cycle and lirilumab 240 mg IV every 4 weeks until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 24 months.
  Interventions: Drug: Epacadostat; Drug: Nivolumab; Drug: Lirilumab
- Phase 2: Dose Expansion: Treatment Group A: Cohort A1 (Experimental): Participants with unresectable or metastatic melanoma (MEL) were planned to be included in this cohort, who did not receive prior systemic therapy for advanced or metastatic disease to receive epacadostat in combination with nivolumab and ipilimumab at the MTD/PAD determined from dose escalation phase.
  Interventions: Drug: Epacadostat; Drug: Nivolumab; Drug: Ipilimumab
- Phase 2: Dose Expansion: Treatment Group A: Cohort A2 (Experimental): Participants with advanced or metastatic non-small cell lung cancer (NSCLC) were planned to be included in this cohort, who have received no more than 1 prior line of platinum-based chemotherapy for advanced or metastatic disease to receive epacadostat in combination with nivolumab and ipilimumab at the MTD/PAD determined from dose escalation phase.
  Interventions: Drug: Epacadostat; Drug: Nivolumab; Drug: Ipilimumab
- Phase 2: Dose Expansion: Treatment Group B: Cohort B1 (Experimental): Participants with recurrent or metastatic serotonin norepinephrine reuptake inhibitor (SCCHN) were planned to be included in this cohort, who received no more than 1 prior line of platinum-based chemotherapy for recurrent or metastatic disease to receive epacadostat in combination with nivolumab and lirilumab at the MTD/PAD determined from dose escalation phase.
  Interventions: Drug: Epacadostat; Drug: Nivolumab; Drug: Lirilumab

INTERVENTIONS:
Drug: Epacadostat — Phase 1: Epacadostat at the protocol-defined dose twice daily. Phase 2: Epacadostat at the recommended dose from Phase 1.
  Other Names: INCB024360
Drug: Nivolumab — Nivolumab at the protocol-specified dose and schedule.
  Other Names: Opdivo®; BMS-936558
Drug: Ipilimumab — Ipilimumab at the protocol-specified dose and schedule.
  Other Names: Yervoy®; BMS-734016
  Arms: Phase 1: Dose Escalation: Treatment Group A: Cohort 1 Epacadostat 50 mg BID; Phase 1: Dose Escalation: Treatment Group A: Cohort 2 Epacadostat 100 mg BID; Phase 2: Dose Expansion: Treatment Group A: Cohort A1; Phase 2: Dose Expansion: Treatment Group A: Cohort A2
Drug: Lirilumab — Lirilumab at the protocol-specified dose and schedule.
  Other Names: IPH2102; BMS-986015
  Arms: Phase 1: Dose Escalation: Treatment Group B: Cohort 1 Epacadostat 50 mg BID; Phase 1: Dose Escalation: Treatment Group B: Cohort 2 Epacadostat 100 mg BID; Phase 2: Dose Expansion: Treatment Group B: Cohort B1

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and efficacy of epacadostat when given in combination with nivolumab and ipilimumab, and in combination with nivolumab and lirilumab, in participant with advanced or metastatic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* During Phase 1, participant with locally advanced or metastatic solid tumors with disease progression on or after treatment with available therapies, or who are intolerant to treatment, or who refuse standard treatment.
* During Phase 2, participant with advanced cancer who have received at least one prior therapy or are treatment naive, depending on the specified tumor type.
* Presence of measurable disease per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Expected survival of ≥ 12 weeks.

Exclusion Criteria:

* Laboratory and medical history parameters not within the Protocol-defined range.
* Receipt of anticancer medications or investigational drugs within Protocol-defined time frames.
* Previous radiotherapy within 7 days of Cycle 1 Day 1.
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Prior treatment with any immune checkpoint inhibitor and/or an IDO inhibitor.
* Active infection requiring systemic therapy.
* Any active or inactive autoimmune disease or syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Consultant for Incyte, Study Director — Incyte Corporation
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 4 study centers in the United States from 21 March 2018 to 29 January 2021.
Pre-assignment Details: Participants were to be enrolled in Phase 1: Dose escalation Phase which consisted of 2 Treatment Groups: A (epacadostat, nivolumab, ipilimumab) and B (epacadostat, nivolumab and lirilumab), followed by Phase 2: a tumor-specific cohort Dose expansion Phase, which was to begin when maximum tolerated dose (MTD)/pharmacologically active dose (PAD) of epacadostat was determined in Phase 1. However, the study was terminated prior to enrollment in Phase 1: Treatment Group B and Phase 2 cohorts.
Groups:
- Phase 1: Dose Escalataion: Treatment Group A: Cohort 1 Epacadostat 50 mg BID: Participants with advanced or metastatic solid tumor who have received no more than 2 prior treatment regimens received epacadostat 50 mg BID orally in combination with nivolumab 240 mg on day 1 of each 14 day cycle and ipilimumab 1 mg/kg intravenous (IV) every 6 weeks thereafter on Day 1 of every third treatment cycle until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 24 months.
Period: Overall Study
Arm/Group | Phase 1: Dose Escalataion: Treatment Group A: Cohort 1 Epacadostat 50 mg BID | Phase 1: Dose Escalation: Treatment Group A: Cohort 2 Epacadostat 100 mg BID | Phase 1: Dose Escalation: Treatment Group B: Cohort 1 Epacadostat 50 mg BID | Phase 1: Dose Escalation: Treatment Group B: Cohort 2 Epacadostat 100 mg BID | Phase 2: Dose Expansion: Treatment Group A: Cohort A1 | Phase 2: Dose Expansion: Treatment Group A: Cohort A2 | Phase 2: Dose Expansion: Treatment Group B: Cohort B1
Started | 5 | 6 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 3 | 4 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants enrolled in the study who received at least 1 dose of combination therapy.
Groups:
- Phase 1: Dose Esclataion: Treatment Group A: Cohort 2 Epacadostat 100 mg BID: Participants with advanced or metastatic solid tumor who have received no more than 2 prior treatment regimens received epacadostat 100 mg BID orally in combination with nivolumab 240 mg on day 1 of each 14 day cycle and ipilimumab 1 mg/kg intravenous (IV) every 6 weeks thereafter on Day 1 of every third treatment cycle until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 24 months.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Dose Escalation: Treatment Group A: Cohort 1 Epacadostat 50 mg BID | Phase 1: Dose Esclataion: Treatment Group A: Cohort 2 Epacadostat 100 mg BID | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (8.79) | 53.8 (8.57) | 59.1 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 90.464 (16.3665) | 81.255 (26.5702) | 85.441 (21.9832)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 173.2 (9.20) | 174.2 (3.25) | 173.7 (6.28)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Percentage of Participants With At Least One Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE is any AE either reported for the first time or worsening of a pre-existing event after first dose of study treatment. AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurs after a participant provides informed consent.
Time Frame: Screening through up to 100 days after end of treatment, up to approximately 24 months
Population: Safety population included all participants enrolled in the study who received at least 1 dose of combination therapy. Treatment group B was excluded from this analysis as no participants were enrolled.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Dose Escalation: Treatment Group A: Cohort 1 Epacadostat 50 mg BID | Phase 1: Dose Esclataion: Treatment Group A: Cohort 2 Epacadostat 100 mg BID
Number analyzed (Participants) | 5 | 6
percentage of participants | 100 | 100

2. Primary Outcome: Phase 2: Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: ORR was defined as the percentage of participants with confirmed objective response (OR). Confirmed OR is defined as complete response (CR) or partial response (PR) on two consecutive occasions ≥ 4 weeks apart, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Every 8 weeks for the first 12 months and then every 12 weeks thereafter up to end of treatment (Up to Month 24)
Population: As the study was terminated early due to business decision, with lack of enrollment, the data for this outcome measure was not collected and analyzed as planned.
Arm/Group | Phase 2: Dose Expansion: Treatment Group A: Cohort A1 | Phase 2: Dose Expansion: Treatment Group A: Cohort A2 | Phase 2: Dose Expansion: Treatment Group B: Cohort B1
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Phase 1: Objective Response Rate (ORR) Based on RECIST v1.1
Description: as for outcome 2
Time Frame: Every 8 weeks for the first 12 months and then every 12 weeks thereafter up to end of treatment (Up to Month 24)
Population: as for outcome 2
Arm/Group | Phase 1: Dose Escalation: Treatment Group A: Cohort 1 Epacadostat 50 mg BID | Phase 1: Dose Escalation: Treatment Group A: Cohort 2 Epacadostat 100 mg BID
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Phase 1: Duration of Response (DOR)
Description: DOR was defined as the time from the earliest date of CR or PR until the earliest date at which progression criteria are met as determined by investigator evaluation of radiographic disease assessment per RECIST v1.1, or date of death due to any cause. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline; or the appearance of one or more new lesions.
Time Frame: Every 8 weeks for the first 12 months and then every 12 weeks thereafter up to end of treatment (Up to Month 24)
Population: as for outcome 2
Arm/Group | Phase 1: Dose Escalation: Treatment Group A: Cohort 1 Epacadostat 50 mg BID | Phase 1: Dose Escalation: Treatment Group A: Cohort 2 Epacadostat 100 mg BID
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Phase 1: Progression-free Survival (PFS)
Description: PFS was defined as the time from the start of combination therapy until the earliest date at which progression criteria are met as determined by investigator evaluation of radiographic disease assessment per RECIST v1.1, or date of death due to any cause. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline; or the appearance of one or more new lesions.
Time Frame: Every 8 weeks for the first 12 months and then every 12 weeks thereafter up to end of treatment (Up to Month 24)
Population: as for outcome 2
Arm/Group | Phase 1: Dose Escalation: Treatment Group A: Cohort 1 Epacadostat 50 mg BID | Phase 1: Dose Esclataion: Treatment Group A: Cohort 2 Epacadostat 100 mg BID
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: as for outcome 4
Time Frame: Every 8 weeks for the first 12 months and then every 12 weeks thereafter up to end of treatment (Up to Month 24)
Population: as for outcome 2
Arm/Group | Phase 2: Dose Expansion: Treatment Group A: Cohort A1 | Phase 2: Dose Expansion: Treatment Group A: Cohort A2 | Phase 2: Dose Expansion: Treatment Group B: Cohort B1
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: as for outcome 5
Time Frame: Every 8 weeks for the first 12 months and then every 12 weeks thereafter up to end of treatment (Up to Month 24)
Population: as for outcome 2
Arm/Group | Phase 2: Dose Expansion: Treatment Group A: Cohort A1 | Phase 2: Dose Expansion: Treatment Group A: Cohort A2 | Phase 2: Dose Expansion: Treatment Group B: Cohort B1
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Phase 2: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE was any AE either reported for the first time or worsening of a pre-existing event after first dose of study treatment. AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurs after a participant provides informed consent.
Time Frame: Screening through up to 100 days for treatment Group A and 150 days for treatment Group B after end of treatment, up to approximately 24 months
Population: as for outcome 2
Arm/Group | Phase 2: Dose Expansion: Treatment Group A: Cohort A1 | Phase 2: Dose Expansion: Treatment Group A: Cohort A2 | Phase 2: Dose Expansion: Treatment Group B: Cohort B1
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening through up to 100 days after end of treatment, up to approximately 24 months
Description: Safety population included all participants enrolled in the study who received at least 1 dose of combination therapy.
Groups:
- Total: Total
Arm/Group | Phase 1: Dose Escalation: Treatment Group A: Cohort 1 Epacadostat 50 mg BID | Phase 1: Dose Esclataion: Treatment Group A: Cohort 2 Epacadostat 100 mg BID | Total
All-Cause Mortality (participants affected / at risk) | 1/5 | 2/6 | 3/11
Serious Adverse Events (participants affected / at risk) | 2/5 | 3/6 | 5/11
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Escalation: Treatment Group A: Cohort 1 Epacadostat 50 mg BID (N=5) | Phase 1: Dose Esclataion: Treatment Group A: Cohort 2 Epacadostat 100 mg BID (N=6) | Total (N=11)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Escalation: Treatment Group A: Cohort 1 Epacadostat 50 mg BID (N=5) | Phase 1: Dose Esclataion: Treatment Group A: Cohort 2 Epacadostat 100 mg BID (N=6) | Total (N=11)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (7) | 1 (1) | 4 (8)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 3 (3)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (2) | 4 (4)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 1 (2) | 3 (4)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 3 (4)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT03347123/Prot_SAP_001.pdf